CLINICAL TRIAL: NCT04643977
Title: An Open-Label Uncontrolled Single Center Study for the Evaluation of the Efficacy and Safety of the Dermal Filler "mARG-01-17" in the Facial Rejuvenation Therapy
Brief Title: Assessment of the Safety and Efficacy of the Dermal Filler "mARG-01-17" in Facial Rejuvenation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD/mARG-06-04-2018
Record Dates: First submitted 2020-02-20; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Facial Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesohyal ARGIBENONE (Experimental): Name of the investigation medical device: mesohyal ARGIBENONE Code of the MD for the purpose of the clinical investigation: mARG-01-17 GMDN code: 59131 mARG-01-17 is a dermal filler recommended for cutaneous filling, facial wrinkle improvement and general condition of the skin, which is administered by intradermal injections. It encourages repair and restructuring of skin tissue, reducing the signs of aging.
  Interventions: Device: mARG-01-17 (mesohyal AGRIBENONE)

INTERVENTIONS:
Device: mARG-01-17 (mesohyal AGRIBENONE) — Dermal Filler

SUMMARY:
The aim of the clinical investigation is to evaluate the performance of the mARG-01-17 dermal filler in the context of its efficacy and safety.

DETAILED DESCRIPTION:
The study is an open-label uncontrolled single-center study for the evaluation of the Performance (efficacy and safety) of the dermal filler "mARG-01-17" in the facial rejuvenation therapy. The design is of a not blinded, not randomized, single group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects;
* Age between ≥35 and ≤65 years;
* Subjects with WSRS (Wrinkle Severity Ranking Scale) score between 2 and 3;
* Skin phototype I - VI;
* Subjects with Glogau score between I and III;
* Subjects with either chrono and photoaging wrinkles, wrinkles of expression (Line of expression); Dry and dehydrated skin;
* Subjects who are willing to abstain from any cosmetic or surgical procedures (including botox injection) in the treatment area during the clinical investigation;
* Clinically and anamnestically healthy individual, especially absence of diseases that could interfere with the cutaneous aging evaluation;
* Absence of a history of significant hypersensitivity to food and drugs or known sensitivity to hyaluronic acid;
* Subjects without significant body weight fluctuation;
* Non-smoker and smokers;
* Arterial blood pressure (BP) (after 5 min. at rest in the supine position) systolic 90 - 140 mmHg and diastolic 50 - 90 mmHg;
* Heart rate (HR) (after 5 min. at rest in the supine position) over 50 beats/min and less than 90 beats/min;
* Respiratory rate between 12 - 24 breaths/min;
* Axillar body temperature of up to 370С;
* Clinical-laboratory examinations within the reference ranges or with no clinically significant abnormalities;
* Negative AIDS/HIV test;
* Negative pregnancy test for the women with reproductive potential;
* Reliable and acceptable method of contraception for the women of child-bearing potential;
* Signed written Informed Consent Form.

Exclusion Criteria:

* Subjects who had previously received permanent implants on the treated area;
* Subjects who underwent facial surgery or were injected with dermal fillers in the facial area within the previous 6 months before enrollment;
* Subjects who underwent facial procedures such as laser therapy, chemical peeling, dermo-abrasive treatments, or botulinum toxin injection within 12 months before enrollment;
* Subjects who indicate signs of dermatological problems, such as cutaneous lesions, acne and/or other inflammatory diseases in active phase, hypertrophic scars or a tendency to keloid formation;
* Subjects suffering from systemic diseases or alterations, such as diabetes mellitus, connective tissue diseases, uncontrolled systemic diseases;
* Subjects, suffering from or who have history of immune system disorders, such as autoimmune diseases, HIV positive status, history of immune system degradation or recurrent herpes simplex or who are undergoing treatment with immunosuppressors or immunotherapy;
* Subjects with known allergy or hypersensitivity to salicylic acid or its derivatives, any of the components of the product or cosmetic fillers to hyaluronic acid;
* Pregnant women;
* Breastfeeding women;
* Absence of a reliable and effective method of contraception;
* Subjects who are currently receiving another investigational treatment or who had participated in another clinical investigation within 30 days prior to study enrollment;
* Subjects who suffer from another medical condition or who are receiving medication that in the Principal Investigator's judgment would prohibit inclusion in the study;
* Subjects with limited mental activity and consistent comprehension ability; sportsmen and individuals on strenuous physical loading; prisoners;
* Refusal to sign the Informed Consent Form.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
The absolute change in Global Aesthetic Improvement Scale (GAIS) | Between Day 0 to Day 90 (up to 12 weeks)
  A 5-point scale rating global aesthetic improvement in appearance, compared to pre-treatment, as judged by the Principal Investigator. Grade 1 - Exceptional improvement, grade 5 - Worsened.
Safety endpoint | Between Day 0 to Day 90
  The frequency and severity of adverse events (AEs)

SECONDARY OUTCOMES:
The absolute change in Global Aesthetic Improvement Scale (GAIS) | Between Day 0 and Days 15, 30, 45, 60 (up to 2, 4, 6 and 8 weeks respectively)
  A 5-point scale rating global aesthetic improvement in appearance, compared to pre-treatment, as judged by the Principal Investigator. Grade 1 - Exceptional improvement, grade 5 - Worsened.
The change in Wrinkle Severity Ranking Scale (WSRS) | Between Day 0 and Days 15, 30, 45, 60 and 90 (up to 2, 4, 6, 8 and 12 weeks respectively)
  A validated five-point reference scale with photographs for evaluation of the skin condition that classifies deep facial wrinkles, like the nasolabial folds. as judged by the Principal Investigator.Grade 1 - the Best result, grade 5 - being the worst result.
Subject satisfaction | Days 15, 30, 45, 60 and 90 (up to 2, 4, 6, 8 and 12 weeks respectively)
  A subject questionnaire including 5 point scale to evaluate the participant's satisfaction - 1 being very much improved and 5 - worsened.

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Bayateva, MD, Principal Investigator — Medical Center Asklepii" OOD
Locations (1):
- "Medical Center Asklepii" OOD, Dupnitsa, Bulgaria

IPD SHARING:
Plan to Share IPD: No